CLINICAL TRIAL: NCT06094478
Title: Implementation of a Stroke Protocol for Emergency Evaluation and Disposition
Brief Title: Hospital Implementation of a Stroke Protocol for Emergency Evaluation and Disposition
Acronym: HI-SPEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: University of Miami (Other); Yale University (Other); University of Cincinnati (Other); Weill Medical College of Cornell University (Other); University of Utah (Other); Emory University (Other); University of Michigan (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB22-1932; 1U01NS131797-01 (NIH)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-04

CONDITIONS: Stroke, Acute; Ischemic Stroke, Acute; Hemorrhagic Stroke
Keywords: interhospital transfer; quality improvement; implementation science; stroke systems of care
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, prospective cluster-randomized, controlled study designed to establish the effectiveness of a multi-component DIDO intervention, the HI-SPEED Protocol, to reduce the median DIDO time for acute ischemic stroke (primary outcome) and for hemorrhagic stroke (secondary outcome) and increase the proportion of acute ischemic stroke patients with good functional outcomes after endovascular therapy (secondary outcome), defined as a 3-month modified Rankin Score of 0-2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Phase (No Intervention): Pre-implementation of HI-SPEED Protocol
- Implementation Phase (Active Comparator): Post-Implementation of HI-SPEED Protocol
  Interventions: Behavioral: HI-SPEED Protocol

INTERVENTIONS:
Behavioral: HI-SPEED Protocol — The HI-SPEED Protocol or Bundle consists of 7 components including 1) stroke screening scales, 2) imaging pathways, 3) telestroke operations, 4) a best practice alert, 5) stroke team communication tool, 6) door-to-needle (thrombolysis) treatment pathway, and 7) a standardized hand-off tool. This protocol will be implemented at each participating health system in clusters of 2 health systems.
  Other Names: HI-SPEED Bundle
  Arms: Implementation Phase

SUMMARY:
Most stroke patients are initially evaluated at the closest hospital but some need to be transferred to a hospital that can provide more advanced care. The "Door-In-Door-Out" (DIDO) process at the first hospital can take time making transferred patients no longer able to get the advanced treatments. This study will help hospitals across the US "stand up" new ways to evaluate stroke patients, decide who needs to be transferred, and transfer them quickly for advanced treatment.

DETAILED DESCRIPTION:
Nearly 800,000 people in the United States (US) each year experience acute stroke, which remains the leading cause of adult disability and 5th leading cause of death. Despite the proliferation of stroke centers nationwide, almost half of the US population lives beyond a 60-minute drive of a comprehensive stroke center (CSC) and many patients require inter-hospital transfer (IHT) from a non-CSC to a CSC. Building upon prior work to reduce door-in-door-out (DIDO) time at referring hospitals, this proposal entitled "Hospital Implementation of a Stroke Protocol for Emergency Evaluation and Disposition (HI-SPEED)" study seeks to (1) implement a novel, evidence-based, multi-component DIDO intervention in eight diverse stroke systems of care across multiple regions of the US and (2) conduct a dual evaluation of its effectiveness in reducing median DIDO time (primary outcome) and disability (secondary outcome) and of the fidelity and quality of implementation. The HI-SPEED study will definitively establish the effectiveness and generalizability of a multi-component evidence-based DIDO intervention and provide information about contextual adaptations for high-quality implementation and widespread dissemination. This study benefits from our well-established interdisciplinary expertise in stroke, emergency and prehospital medicine, systems and quality engineering, health services research, and strong multicenter research collaborations. Findings from HI-SPEED will have substantial implications for a wide range of hospitals and stroke systems of care worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Final diagnosis: AIS, ICH, or SAH

Exclusion Criteria:

* Final diagnosis: TIA or stroke NOS
* Age <18 years
* Comfort care measures on day 0 or 1
* Left hospital against medical advice
* Enrolled in clinical trial related to stroke that is competing with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
DIDO time in acute ischemic stroke patients | Baseline
  Time from ED arrival to ED departure prior to transfer to a comprehensive stroke center among ischemic stroke patients

SECONDARY OUTCOMES:
DIDO time in acute hemorrhagic stroke patients | Baseline
  Time from ED arrival to ED departure prior to transfer to a comprehensive stroke center among hemorrhagic stroke patients
Modified Rankin Scale score at 3 months in acute ischemic stroke patients undergoing endovascular therapy | 3 months post-stroke
  Proportion of acute ischemic stroke patients who undergo endovascular therapy and achieve good functional outcome (mRS 0-2) at 3 months post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Prabhakaran, MD, MS, Principal Investigator — University of Chicago; Jane Holl, MD, MPH, Principal Investigator — University of Chicago
Locations (7):
- United States (7):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Jackson Memorial Hospital, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - UChicago Medicine Ingalls Memorial Hospital, Chicago, Illinois
  - New York Presbyterian - Weill Cornell Hospital, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Utah Health, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Only aggregate data and analyses will be shared between sites while sites will have IPD for their own site level data only.

REFERENCES:
- [Background] Anderson CS, Chalmers J, Stapf C. Blood-pressure lowering in acute intracerebral hemorrhage. N Engl J Med. 2013 Sep 26;369(13):1274-5. doi: 10.1056/NEJMc1309586. No abstract available. PMID 24066751
- [Background] Richards CT, Holl JL, Khorzad R, Prabhakaran S. Abstract TMP70: Simulation Modeling Predicts Actual Patient Transport Rates Following the Implementation of a Prehospital Comprehensive Stroke Center DirectTransport Protocol. Stroke. 2020;51(Suppl_1):ATMP70-ATMP70.
- [Background] Menon BK, Saver JL, Goyal M, Nogueira R, Prabhakaran S, Liang L, Xian Y, Hernandez AF, Fonarow GC, Schwamm L, Smith EE. Trends in endovascular therapy and clinical outcomes within the nationwide Get With The Guidelines-Stroke registry. Stroke. 2015 Apr;46(4):989-95. doi: 10.1161/STROKEAHA.114.007542. Epub 2015 Feb 13. PMID 25681065
- [Background] Saver JL, Fonarow GC, Smith EE, Reeves MJ, Grau-Sepulveda MV, Pan W, Olson DM, Hernandez AF, Peterson ED, Schwamm LH. Time to treatment with intravenous tissue plasminogen activator and outcome from acute ischemic stroke. JAMA. 2013 Jun 19;309(23):2480-8. doi: 10.1001/jama.2013.6959. PMID 23780461
- [Background] Mendelson SJ, Aggarwal NT, Richards C, O'Neill K, Holl JL, Prabhakaran S. Racial disparities in refusal of stroke thrombolysis in Chicago. Neurology. 2018 Jan 30;90(5):e359-e364. doi: 10.1212/WNL.0000000000004905. Epub 2018 Jan 3. PMID 29298854
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560